CLINICAL TRIAL: NCT03120585
Title: Multicenter Randomized Controlled Trial Of Restrictive Fluid Management For Respiratory Distress in the Newborn Period
Brief Title: Fluid Restriction in Respiratory Distress of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Universidad Abierta Interamericana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4688
Record Dates: First submitted 2015-09-08; First posted 2017-04-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Respiratory Distress Syndrome, Newborn; fluid restriction
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid Management Intervention (Experimental): Restricting IV fluids to infants with respiratory distress to mimic fluid intake of normal healthy breast fed infants (less fluid that current standard of care)
  Interventions: Other: Fluid Management Intervention
- Control Group (No Intervention): Infants with respiratory distress will receive standard of care fluid management.

INTERVENTIONS:
Other: Fluid Management Intervention — Fluid management intervention is fluid restriction to 60 mL/kg/day on Day of Life (DOL) 1 for preterm and 40 mL/kg/day on DOL 1 for term neonates, calculated as total of IV and enteral fluid intake. Infants randomized to low infusion with be placed on 10% dextrose and the Infant will be monitored by obtaining serum glucose levels by point of care testing. Glucose infusion rates (GIR) would be calculated to the corresponding serum glucose and recorded. After 24 hours, infusion rate will be increased to 60ml/kg/d providing minimum GIR >4mg/kg/d. . Total fluid intake will be increased by 20 mL/kg/day until 150 mL/kg/day .
  Arms: Fluid Management Intervention

SUMMARY:
The object of this study is to determine the best way to care for infants with respiratory distress. The investigators are testing a method of feeding fluids to infants with respiratory distress in amounts similar to what healthy breastfed babies eat when they are feeding on demand, and comparing this method to the current standard of care for feeding fluids to infants with respiratory distress. These methods of feeding fluids to the study infants will continue until the infants are able to feed normally by mouth. The study will include about 400 infants across five sites in the United States, Chile and Argentina.

DETAILED DESCRIPTION:
Infants with respiratory distress syndrome will be enrolled within the first twelve hours of life, and randomly assigned to one of two groups: the first group will receive the interventional fluid management method, and the second (the control group) will receive the current standard of care for fluid management. To standardize respiratory care across all five study sites, a computer-based algorithm for respiratory support management based on objective markers of respiratory distress will guide clinician management decisions. However, each infant's medical team will make all final decisions on respiratory treatment and IV fluid management. Any study infant who experiences dehydration and/or low blood sugar during the course of the study will be removed from the study and be treated for the condition.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born between 34-0/7 and 41-6/7 weeks gestational age (GA) at birth with primary pulmonary disease of the newborn including Transient Tachypnea of the Newborn (TTN), Respiratory Distress Syndrome (RDS), air leak syndrome, pneumonia, or meconium aspiration syndrome in the first 12 hours of life will be eligible for inclusion in this study.
* Those neonates who are intubated for administration of exogenous surfactant but who are immediately extubated to non-invasive respiratory support after surfactant administration will remain eligible for study inclusion.

Exclusion Criteria:

* Neonates with a genetic abnormality or congenital anatomic anomaly

Subsequent Study Exclusion resulting in removal from study:

* Neonates who subsequently undergo endotracheal intubation and mechanical ventilation for refractory respiratory distress
* Neonates with hypoglycemia or clinical evidence of dehydration or volume depletion requiring fluid bolus
* Infants that are transported out of the participating site prior to study endpoint.

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Time from birth to first oral feeding | every 24 hours for up to 168 hours
  Total Hours until first oral feeding

SECONDARY OUTCOMES:
Duration of Respiratory Support | every 3 hours for up to 168 hours
  Total hours of Respiratory Support
Total Duration of NICU stay | every 24 hours up to 12 weeks
  Length of Stay in the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Makkar, MD, Study Director — University of Oklahoma HSC
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Comanche county Memorial hospital, Lawton, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bell EF, Acarregui MJ. Restricted versus liberal water intake for preventing morbidity and mortality in preterm infants. Cochrane Database Syst Rev. 2014;2014(12):CD000503. doi: 10.1002/14651858.CD000503.pub3. Epub 2014 Dec 4. PMID 25473815
- [Background] Stroustrup A, Trasande L, Holzman IR. Randomized controlled trial of restrictive fluid management in transient tachypnea of the newborn. J Pediatr. 2012 Jan;160(1):38-43.e1. doi: 10.1016/j.jpeds.2011.06.027. Epub 2011 Aug 11. PMID 21839467